CLINICAL TRIAL: NCT02960607
Title: A Phase II Study of High-dose Icotinib in Previously Treated Non-small Cell Lung Cancer Patients With Epidermal Growth Factor Receptor Mutation
Brief Title: High-dose Icotinib Treatment Beyond Progression in EGFR Mutant NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Yutao Liu, Associate Chief Physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-L-059
Record Dates: First submitted 2016-11-08; First posted 2016-11-09 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib

ARMS (1):
- Icotinib (Experimental): 250mg, tid until disease progression or unacceptable toxicities occurred
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Icotinib (250mg tid) until disease progression or unacceptable toxicities occurred.

SUMMARY:
The purpose of this study is to investigate whether high-dose icotinib treatment beyond disease progression is beneficial for NSCLC patients who have EGFR mutation and who have responded to EGFR TKI.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IIIB/IV NSCLC
* Investigator confirmed progression according RECIST 1.1 during previous icotinib treatment
* Patients whose tumors:

  * are EGFR mutation-positive or
  * T790M mutation-negative
* Performance status: WHO 0-2
* Measurable disease according to RECIST 1.1

  * at least one measureable lesion .if only one measureable lesion, the biological nature must be confirmed by cytology or histology
  * a single diameter of lesion could be measured by at least one of the following methods: Chest or abdominal computed tomography(CT)or magnetic resonance imaging(MRI),conventional methods of diameter at least 20mm diameter spiral CT OR at least 10mm
* ANC ≥ 1.5*109/L, Platelets ≥ 75*109/L, Hgb≥ 9g/dL, Alanine amino transferase ≤ 2 × Upper limit of normal (ULN), Alkaline phosphatase ≤ 2.5 × ULN (< 5 × ULN if liver metastases), Serum Creatinine ≤ 1.5 × ULN
* Women of childbearing age must have a pregnancy test 7 days before treatment and the result were negative ,men of childbearing age: surgical sterilization or treatment during and after the end of three months to take contraceptive measures
* Patient must be able to comply with the protocol

Exclusion Criteria:

* Patient with symptomatic central nervous system metastases
* Patient has known active hepatitis B or C, or HIV infection
* Pregnant or breastfeeding.
* Patient with uncontrolled undercurrent illness or circumstances that could limit compliance with the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences, Beijing, China